CLINICAL TRIAL: NCT03949972
Title: The FOrMe Registry (The German Focal Segmental Glomerulosclerosis and Minimal Change Disease Registry)
Acronym: FOrMe
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Paul Brinkkoetter (Other)
Collaborators: German Research Foundation (Other); Medical Faculty and the Faculty of Natural Sciences of the University of Cologne (Unknown); Cluster of Excellence on Cellular Stress Responses in Ageing-Associated Diseases (Unknown); Cologne Center for Genomics (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Paul Brinkkoetter, Consultant in Nephrology, Scientific Coordinator KFO 329, University of Cologne
Organization: University of Cologne (Other)
Other Study IDs: 005
Record Dates: First submitted 2018-12-03; First posted 2019-05-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Glomerulosclerosis, Focal Segmental; Minimal Change Disease; Idiopathic Nephrotic Syndrome
Keywords: Focal and Segmental Glomerulosclerosis; Focal & Segmental Glomerulosclerosis; FSGS; Minimal change disease; MCD; Nephrotic Syndrome
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Macular dystrophy, corneal type 1; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Blood (plasma, serum), urine, DNA, feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A - Pediatric Cohort: Pediatric patients until 18 years of age presenting with or diagnosed with idiopathic nephrotic syndrome or a biopsy-proven diagnosis of MCD or FSGS.
  Interventions: Other: Biosampling
- B -Adult Cohort: Adult patients 18 years and above with a biopsy-proven diagnosis of primary or secondary FSGS or MCD.
  Interventions: Other: Biosampling

INTERVENTIONS:
Other: Biosampling — Biosampling at initial visit and follow-up visits

SUMMARY:
In a monocentric, later multicentric prospective approach the FOrMe registry (The German Focal Segmental Glomerulosclerosis and Minimal Change Disease Registry) aims to generate a longitudinal cohort of 150 pediatric cases of idiopathic nephrotic syndrome and 350 adult cases of biopsy-proven Minimal Change Disease (MCD) or Focal and Segmental Glomerular Sclerosis (FSGS) over 10 years. The registry will provide a repository for biomaterials such as blood samples, DNA, urine, feces, and tissue biopsies that will be accessible to collaborators to facilitate future research on pathogenesis, diagnostics, and treatment.

DETAILED DESCRIPTION:
Idiopathic Nephrotic Syndrome is characterized by proteinuria, volume retention, hyperlipidemia, hypoalbuminemia. As Minimal Change Disease (MCD) represents by far the most prevalent underlying diagnosis in children older than 1 year, a kidney biopsy is usually deferred in these cases. In adolescence and adults, a kidney biopsy is crucial for the diagnosis because MCD and FSGS account for only 10-15 and 12-35 percent of all cases of nephrotic syndrome respectively. Pathomechanisms as well as optimal treatment remain elusive as systematic trials are scarce and hampered by low incidence and heterogenicity of the clinical presentation. To bridge this informational gap, the investigators identified the need for a German registry of pediatric and adult patients with idiopathic nephrotic syndrome (in children) and biopsy-proven MCD/FSGS (in adults).

The registry will record clinical data of participants regarding basic demographics, initial presentation, hereditary traits, disease course and treatment modalities as well as quality of life, concomitant diseases, and comedication. During the initial visit and to a lesser intent on follow-up visits, biomaterials (blood, urine, DNA, feces, tissue) will be collected and stored in a state-of-the art biobank. This material will be available to collaborators to support research on idiopathic nephrotic syndrome and MCD/FSGS. By the time of completion, the registry will provide data on clinical courses and outcome of approximately 500 patients that can easily be correlated with biomaterials giving insight into risk factors, prognostic parameters, and association with comorbidities.

Tissue sections of all patients that undergo kidney biopsy (all adult and some pediatric patients) will be digitalized, annotated, and analyzed by a panel of nephropathologists. Histopathologic features will be individually assessed and scored according to a set of descriptors that was developed and is used by the American NEPTUNE (Nephrotic Syndrome Study Network).

ELIGIBILITY:
Inclusion Criteria (cohort A):

* written informed consent
* 17 or less years of age
* idiopathic nephrotic syndrome

Inclusion Criteria (cohort B):

* written informed consent
* older or equal to 18 years of age
* biopsy-proven primary or secondary FSGS or MCD or biopsy-proven recurrence of disease in kidney transplant.

Exclusion Criteria (both cohorts):

* Prior kidney transplant without biopsy-proven recurrence
* A clinical diagnosis of other glomerular disease resulting in secondary MCD or FSGS as judged by the treating physicians.
* Refusal to provide written informed consent
* (Anticipated) incompliance with visit schedule

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients until 18 years of age presenting with or diagnosed with idiopathic nephrotic syndrome or a biopsy-proven diagnosis of MCD or FSGS. Candidate participants need to be willing to provide written informed consent.
  Adult patients 18 years and above with a biopsy-proven diagnosis of primary or secondary FSGS or MCD. Candidate participants need to be willing to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Average Annual Change in estimated glomerular filtration rate (eGFR) | 5-15 years
  Outcome measure: eGFR loss in ml/min/year. Higher values are considered worse outcome.
Incidence of End-stage Renal Disease (ESRD) | 5-15 years
  Documented initiation of chronic renal replacement therapy regardless of type.
Incidence of Death | 5-15 years
  Documented patient death due to any cause
Incidence of Kidney Transplantation | 5-15 years
  Documented kidney transplantation regardless of type (living donor, cadaveric donor)
Changes in Quality of Life (adults patients) | 5-15 years
  Patient-reported outcome will be assessed using Quality of Life questionnaires at regular intervals using the SF-36 questionnaire.
  For reference see https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html The SF-36 questionnaire measures eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. All items are scored so that a high score defines a more favorable health state. Lowest and highest possible scores are 0 and 100. Scores represent the percentage of total possible score achieved.
  Original publication: Ware, J.E., Jr., & Sherbourne, C.D. "The MOS 36-Item Short-Form Health Survey (SF-36): I. Conceptual Framework and Item Selection,". Medical Care, 30:473-483, 1992.
Changes in Quality of Life (pediatric patients) | 5-15 years
  Patient-reported outcome will be assessed using Quality of Life questionnaires at regular intervals using the PedsQL questionnaire.
  For reference see https://www.pedsql.org/score.html The PedSQL questionnaire measures four health concepts: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life). To create Scale Scores, the mean is computed as the sum of the items over the number of items answered (this accounts for missing data). To create the Total Scale Score, the mean is computed as the sum of all the items over the number of items answered on all the Scales.

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Brinkkoetter, MD, Study Director — University Hospital of Cologne, Cologne, Germany
Locations (12):
- Germany (12):
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Uniklinik RWTH Aachen, Aachen
  - Charité University Hospital, Berlin
  - Kindernierenzentrum Bonn, Bonn
  - Kindernephrologie Dachau, Dachau
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - University Hospital Heidelberg, Heidelberg
  - Klinikum St. Georg, Leipzig
  - University Hospital Marburg, Marburg
  - University Hospital Münster, Münster
  - Klinikum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: Yes
Biosamples as well as patient data will be available to collaborators after revision of research application by a steering committee.
Time Frame: 5-15 years
Access Criteria: Actively contributing to registry and approval by international steering committee.

REFERENCES:
- [Derived] Osterholt T, Todorova P, Kuhne L, Ehren R, Weber LT, Grundmann F, Benzing T, Brinkkotter PT, Volker LA. Repetitive administration of rituximab can achieve and maintain clinical remission in patients with MCD or FSGS. Sci Rep. 2023 Apr 28;13(1):6980. doi: 10.1038/s41598-023-32576-7. PMID 37117201
- See also: CRU 329 Homepage — http://www.podocyte.org